CLINICAL TRIAL: NCT01699516
Title: A Prospective Study on Qualitative and Quantitative Non-invasive Evaluation of Intestinal Acute Graft-vs-host Disease by Contrast Enhanced Ultrasound Sonography
Brief Title: Non-invasive Contrast Enhanced Ultrasound Sonography in Intestinal Acute Graft-vs-Host Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Dr Edoardo Benedetti, MD, University of Pisa
Other Study IDs: IRB33982
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Intestinal GVHD; Neutropenic Enterocolitis
Keywords: allogeneic transplantation; intestinal graft-vs.-host disease; contrast enhanced ultrasound sonography
MeSH Terms: conditions — Enterocolitis, Neutropenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intestinal graft vs host disease: Patients with biopsy-proven intestinal acute GVHD in the setting of an allogenic transplant
- Control group: In the setting of an allogenic bone marrow transplant: patients with biopsy-proven stomach GVHD without intestinal symptoms and patients with neutropenic enterocolitis. Normal volunteers.

SUMMARY:
Intestinal acute graft-vs-host disease (GVHD) is a life-threatening complication after allogeneic hematopoietic cell transplantation. Non-invasive diagnostic procedures are still lacking and diagnosis is difficult. We hypothesized that contrast-enhanced ultrasound sonography (CEUS) could detect microcirculation changes of the bowel walls during intestinal GVHD and help to detect and monitor treatment response. We employed CEUS to prospectively evaluate intestinal GVHD in 83 consecutive transplant patients between 2008 and 2011. Fourteen /83 patients with biopsy-proven intestinal GVHD were selected as study group. Fourteen patients with biopsy-proven stomach GVHD without intestinal symptoms (N=16), normal volunteers (N=6) and patients with neutropenic enterocolitis (N=4), were chosen as control group. All patients were evaluated with both standard transabdominal ultrasonography (US) and CEUS at the onset of intestinal symptoms, during clinical follow up and at flare of symptoms. Standard US revealed non-specific bowel wall thickening, and simultaneous involvement of multiple intestinal segments in 9/14 patients. CEUS showed three distinct patterns of microcirculation changes that correlated with GVHD activity. These findings were not observed in the control group. Moreover, CEUS findings correlated with treatment response and predicted flare of intestinal symptoms. CEUS is a non-invasive, easily reproducible bed-side tool to detect and monitor intestinal GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Bone Marrow Transplant
* intestinal acute graft versus host disease
* stomach GVHD
* neutropenic enterocolitis

Exclusion Criteria:

no biopsy proven intestinal or stomach GVHD no neutropenic enterocolitis

Ages: 22 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the setting of allogenic transplant: intestinal acute graft vs host disease (GVHD), stomach GVHD, neutropenic enterocolitis.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Chiara Hospital University of Pisa, Pisa, Italy